CLINICAL TRIAL: NCT03763006
Title: Comparison in the Efficiency and Safety Between the Applications of New Hypochlorous Acid Eyelid Wipes and Povidone Lodine on the Eye Surface
Brief Title: Efficacy and Safety of Ocudox Lid Wipes Compared to Traditional Lid Cleaning
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Senior Consultant, Singapore National Eye Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R1451/34/2017; 2017/2387 (Registry Identifier: SingHealth CIRB)
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2018-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Ocudox lid wipes
Who Masked: Investigator
Masking Description: Investigator will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ocudox lid wiped (Experimental)
  Interventions: Procedure: Eyelid cleaning
- Povidone Iodine (Active Comparator)
  Interventions: Procedure: Eyelid cleaning

INTERVENTIONS:
Procedure: Eyelid cleaning — This is a pure hypochlorous acid that kills many microbes, but remain very friendly and non-toxic for the ocular surface.

SUMMARY:
The use of povidone iodine solution for prophylaxis of endophthalmitis is well established for intraocular procedures like cataract surgery and for injections of anti-VEGF agents for retinal diseases such as age-related macular degeneration. Unfortunately iodine is unfriendly to the ocular surface, and when repeated often enough (some patients require up to monthly injections of anti-VEGF agents for the entire year), corneal epitheliopathy and secondary dry eye results. Unfortunately, there is no good alternative to cleaning patient's eyelid at the moment. Ocudox is a relatively new antibacterial product (spraying on eyelid wipe) which contains Neutrox (pure hypochlorous acid) that kills many microbes, but remain very friendly and non-toxic for the ocular surface.

DETAILED DESCRIPTION:
In a multicentre study involving 71 eyes, reported at a conference abstract (ARVO), Avenova (similar ingredients as Ocudox) reduces bacteria on ocular skin surface by more than 90% without altering the diversity of bacteria on the ocular skin surface in any significant way. This lowering of the bacterial load was particularly noteworthy for all staphylococci, including S. epidermidis, the most frequently recovered species. At 20 minutes following treatment, 138 unique bacterial strains belonging to 26 different species were recovered.

However, the efficacy of anti-microbial action has not been compared to the gold standard of a single wipe with povidone iodine solution. Investigator intend to compare pre and post treatment of Ocudox and a single use of povidine iodine solution at Day 14 in terms of the alteration of the conjunctival microbiome of the eye and the effect on the ocular surface.

Clinical significance The study has implications on the prophylaxis of infection in many common ophthalmic procedures conducted in Singapore National Eye Centre and many places in the world.

1. OBJECTIVES The aim of this study is to compare pre and post-treatment of the application of Ocudox to a single use of povidine iodine solution at Day 14in terms of the alteration of the conjunctival microbiome and the integrity of the eye.
2. EXPECTED RIKS AND BENEFITS There would be no expected risk involved as all the evaluations are non-invasive. However, there will be some slight discomfort from measure tear volume or tear collection (Schirmer's strips) and also slight discomfort from culturing procedure.

There are no known benefits from participation in this study. However, this project may have the potential to prevent infection in many common ophthalmic procedures conducted in Singapore National Eye Centre and many places in the world.

3. STUDY POPULATION 3.1. List the number and nature of subjects to be enrolled. Due to the nature of the preliminary study, six participants with Meibomian Gland Dysfunction (MGD) will be recruited from Singapore National Eye Centre. Participants will be randomised into either Ocudox group or single use povidine iodine solution.

n= 3 (Ocudox group) n= 3 (Single use povidine iodine solution)

3.2. Criteria for Recruitment and Recruitment Process

1. Participants meet all the inclusion criteria listed below. 2. Clear of exclusion criteria. Permission would be sought from the attending doctors before participants are being recruited.

Eligible participants will be counselled on the study by the study coordinator. If the participant is interested, the study coordinator will then accompany the participant to SERI level 5 for the relevant assessments. Informed written consent will be obtained from all participants.

3.3. Inclusion Criteria Participants must meet all of the inclusion criteria to participate in this study.

1. Participants must be 50 to 60 years old with Meibomian Gland Dysfunction (MGD) 2. Clear of exclusion criteria 3. Willing to perform all eye examinations in this study 3.4. Exclusion Criteria Participants meeting any of the exclusion criteria will be excluded from this study.

1. Participants diagnosed with diabetes
2. No recent eye surgery or eye procedure within 1 month
3. Participants who are unsuitable for Oculus K5M recording such as musculoskeletal problems
4. Participants who are unable to tolerate Oculus K5M recording machine
5. Is pregnant, lactating or planning a pregnancy
6. Any other specified reason as determined by clinical investigator

4. STUDY DESIGN AND PROCEDURES/METHODOLOGY This is a randomised interventional trial with Ocudox eyelid wipes and povidine iodine solution.

Study visits and duration:

Trial arms No. of study visits Study duration Ocudox eyelid wipes 3 21±3 days Povidine iodine solution 3 21±3 days Recruitment duration: One year

Treatment arms and randomisation:

There will be 2 trial arms (parallel groups) in this study:

A. Ocudox eyelid wipes n=3 B. Povidine iodine solution n=3

Randomisation and Blinding

The randomisation procedure used will entail:

1. Presence of two witnesses
2. Drawing of lots
3. Randomization codes for the 2 groups will be noted. For e.g. 001A, 002B, etc.
4. Study information related to randomisation will be filed and kept at SERI
5. Only unblinded personnel have access to the randomization code file

There will be blinded and unblinded study team members in this study. Blinded study team members will only be performing the procedures as described below. Unblinded study team members will dispense the study product, counsel participants on directions for using Ocudox eyelid wipes and also to clean the eyelid and conjunctiva if randomised to Povidone Iodine,

Directions for using Ocudox eyelid wipes:

Participant who received Ocudox eyelid wipes will be instructed to clean the eyelid according to manufacturer's protocol during the study period (twice a day). A diary chart will be given to all participants at the end of baseline visit. Participants will be asked to fill up the diary chart whenever Ocudox eyelid wipes was used.

Directions for cleaning with Povidone Iodine:

• Pour 10ml of 10% Povidone Iodine into a 50ml Falcon tube.

* Dilute 10% of Povidone Iodine to 5% by pouring 10ml of saline and 10ml of Povidone Iodine into a 50ml Falcon tube
* Prepare gauze and dip into the 10% Povidone Iodine solution
* Clean participant's exterior eye at least 2-3 times
* Next, flush the interior of the participant's eye with 5% Povidone Iodine
* Using a pasture pipette, flush the interior of the participant's eye
* Wait for 5 minutes
* After 5 minutes, rinse off with saline solution
* Thereafter, wait for 1 minute before adding tetracaine
* After adding tetracaine, wait for another minute before collection of microbiome swab.

Equipment used:

Oculus Keratograph 5M will be used on the baseline visit and post-treatment visits.

Workflow procedure:

Ocular symptoms will be examined subjectively using standard patient evaluation of eye dryness (SPEED). Oculus Keratograph 5M will be conducted to assess tear meniscal height (TMH), conjunctival redness and Non-invasive Tear Break-Up time (NIKBUT). Meibomain gland evaluator will be used to assess the number of expressible glands. Bacteria on the eye surface will be cultured from one of the conjunctivas (white part of the eyes) and Schirmers I test will carry out to examine tear secretion and tear collection.

Outcomes:

Differences in Tear Meniscus Height, Ocular Redness, Non-invasive Tear Break-up time readings and findings of DNA/RNA between study visits and study groups.

Figure 2. Study workflow

Details of study procedures shown below:

i) SPEED questionnaires Investigator will use the previously validated standard patient evaluation of eye dryness (SPEED) questionnaire, which consists of 2 questions on frequency and severity of dry eye graded on a scale of 0-3 on frequency, and grades 0-4 on severity. Scores from all sub-questions will be added, and the greater the total score (0-28), the more frequent or severe the dry eye (2).

ii) Non-invasive tear break-up time Both Oculus Keratograph 5M (Oculus, Wetzlar, Germany) will be used to perform the non-invasive tear break up time (NIKBUT) (3). Briefly, seated patients blink freely while fixing on a target ahead. Once ready, patients blink twice and then refrain from further blinking. The fully automated instrument will capture any break or distortion in the image of the projected rings on the cornea and the timings will be automatically recorded. One reading will be taken per eye (4).

iii) Conjunctiva redness & Tear meniscus height Oculus Keratograph 5M (Oculus, Wetzlar, Germany) will be used to measure conjunctival redness. After scanning the ocular surface and images captured, grading of the conjunctival hyperemia (0-4) will be automatically performed with subtraction of major conjunctival blood vessels, and temporal bulbar, nasal bulbar and average readings will be obtained. Higher redness scores indicate more hyperemia(5). Height of the tear meniscus can be measured by dragging the ruler option icon and the measured value will appear in mm.

iv) Meibomain Gland Evaluator Meibomian glands will be assessed by gently squeezing the lower eyelids using a device that delivers standardised pressure to the eyelids (Meibomian gland expresser, TearScience, France). Texture of the expressed secretion will be graded as liquid or viscous. The number of expressible glands will be recorded.

v) Collection of microbiome One specimens of microbiome will be collected from both eyes First: a drop of non-preserved tetracaine will be instilled into the conjunctival fornix. After the stinging sensation has resolved, a sterile cotton swap will be used to collect the microbes from the lower conjunctival fornix using a gentle rolling action (up to 8 strokes). The procedure is then repeated for the opposite eye.

These swaps will then be soaked in DNA/RNA Shield (Zymo) reagent and immediately homogenised for 1 minute, stop at 30 seconds, and keep on ice for 1 minute, and homogenized for another 30 seconds. Homogenised samples will be stored at 4°C. This ensures an optimal and sufficient DNA/RNA yield for our purpose. Subsequent nucleic acid extraction, PCR, sequencing, and bioinformatics procedures will be performed by our collaborators. Storage: intended to be analysed within a year, not more than 5 years.

Analysis: Investigator intend to compare composition of known microbes at the specie and genus level after obtaining the reads in the non-human DNA metagenomics signatures.

vi) Schirmers I test Schirmer I test will be done with the standard 5 mm wide Test Strips (Clement Clark) with a notch for folding, without prior anaesthesia. The strips will be positioned over the inferior temporal half of the lower lid margin in both eyes, and participants' eyes will then close. The extent of the wetting will be recorded after 5 minutes, and strips stored at -80˚C until further analysis(7).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 50 to 60 years old with Meibomian Gland Dysfunction (MGD)
2. Clear of exclusion criteria
3. Willing to perform all eye examinations in this study

Exclusion Criteria:

1. Participants diagnosed with diabetes
2. No recent eye surgery or eye procedure within 1 month
3. Participants who are unsuitable for Oculus K5M recording such as musculoskeletal problems
4. Participants who are unable to tolerate Oculus K5M recording machine
5. Is pregnant, lactating or planning a pregnancy
6. Any other specified reason as determined by clinical investigator

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
SPEED Questionnaire | 21 days
  To compare the frequency and severity of dry eye symptoms at baseline and after 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, PhD, Principal Investigator — Singapore Eye Research Institute
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No